CLINICAL TRIAL: NCT03288532
Title: An International Investigator-led Phase III Multi Arm Multi Stage Multi-centre Randomised Controlled Platform Trial of Adjuvant Therapy in Patients With Resected Primary Renal Cell Carcinoma (RCC) at High or Intermediate Risk of Relapse
Brief Title: Renal Adjuvant MultiPle Arm Randomised Trial
Acronym: RAMPART
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: AstraZeneca (Industry); Kidney Cancer UK (Other); Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRC RE06
Record Dates: First submitted 2017-09-04; First posted 2017-09-20 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Renal Cell Carcinoma
Keywords: Renal Cell Carcinoma; Immunotherapy; Multi-Arm Multi-Stage
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — durvalumab; tremelimumab

STUDY DESIGN:
Intervention Model Description: Multi-Arm Multi-Stage Design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A (active monitoring) (No Intervention): Participants randomised to Arm A will be allocated to active monitoring for 1 year, in line with current standard-of-care in resected primary RCC at high or intermediate risk of relapse
- Arm B (durvalumab monotherapy) (Experimental): Participants randomised to Arm B will receive durvalumab (1500mg) 4 weekly for 1 year (13 cycles maximum)
  Interventions: Drug: Durvalumab
- Arm C (durvalumab + tremelimumab) (Experimental): Participants randomised to Arm C will receive durvalumab (administered as per arm B, i.e. 13 cycles maximum) and tremelimumab (75mg) on day 1 and week 4 visits (i.e. 2 cycles)
  Interventions: Drug: Durvalumab; Drug: Tremelimumab

INTERVENTIONS:
Drug: Durvalumab — controlled infusion via an infusion pump into a peripheral or central vein
  Arms: Arm B (durvalumab monotherapy); Arm C (durvalumab + tremelimumab)
Drug: Tremelimumab — controlled infusion via an infusion pump into a peripheral or central vein
  Arms: Arm C (durvalumab + tremelimumab)

SUMMARY:
RATIONALE: The current global standard of care after nephrectomy for localised RCC therefore remains active monitoring (i.e., observation by clinical and radiological means). 30-40% patients with initially localised RCC develop metastatic disease following nephrectomy. Need for adjuvant therapy is most marked in the high risk population where outcomes are predictably poor. However, the risk of recurrence in patients who are of intermediate risk of recurrence is not insignificant. Unfortunately, despite showing efficacy in advanced RCC, the results in the adjuvant setting, so far, are inconclusive.

AIM: RAMPART is a phase III Multi-Arm Multi-Stage randomised controlled platform trial, initiated with three arms. The trial is assessing if durvalumab monotherapy or the combination of durvalumab and tremelimumab can improve Disease Free Survival (DFS) or Overall Survival (OS) compared to the current global standard-of-care (active monitoring). At the start of recruitment, patients with Leibovich scores 3 to 11 will be eligible for randomisation. Accrual of intermediate risk patients (Leibovich scores 3 5) will stop after 3 years or when intermediate risk patients contribute 25% of the total accrual target, whichever is earlier. Recruitment of patients with Leibovich scores 6 to 11 will continue until the accrual target is reached.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven RCC (all cell types of RCC are eligible, except for pure oncocytoma, collecting duct, medullary and transitional cell cancer [TCC]); no evidence of residual macroscopic disease on post-operative CT scan after resection of RCC. Patients with treated bilateral synchronous RCCs are eligible.
2. At the start of recruitment patients with Leibovich score 3-11 will be eligible for randomisation. MRC CTU at UCL will monitor accrual and stop recruiting intermediate risk patients (Leibovich Score 3-5) after three years or when intermediate risk patients contribute 25% of the total accrual target, whichever is earlier. Recruitment of patients with Leibovich Score 6 11 will continue until the accrual target is reached.
3. Patients should have had surgery at least 28 days but no more than 91 days prior to their randomisation date.
4. Post-operative scans should be performed within 28 days prior to randomisation.
5. Patients with microscopically positive resection margins after radical nephrectomy at the nephrectomy bed, renal vein or inferior vena cava are eligible provided the post-operative CT scan shows no evidence of residual macroscopic disease.
6. WHO Performance Status 0 or 1.
7. Patient has archival FFPE pathology tissue available, and agrees to provide at least one sample (FFPE tumour block from nephrectomy, or a minimum of 10 unstained slides), as well as a baseline EDTA blood sample for future translational research).
8. Adequate normal organ and marrow function

   1. Haemoglobin ≥9.0g/dL (transfusions will be allowed within 2 weeks prior to randomisation in order to achieve the entry criteria).
   2. Absolute neutrophil count (ANC) ≥1.5 x 109/L (≥1500 per mm3).
   3. Platelet count ≥100 x 109 (≥100,000 per mm3).
   4. Bilirubin ≤1.5 x ULN (This will not apply to subjects with confirmed Gilbert's syndrome (i.e., persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of haemolysis or hepatic pathology), who will be allowed only in consultation with their physician).
   5. AST/ALT ≤2.5 x ULN.
   6. Calculated Creatinine Clearance level >40mL/min by Cockcroft Gault formula (using actual body weight).
9. 12-lead ECG on which QTcF must be <450 ms. In case of clinically significant ECG abnormalities, including a QTcF value ≥450 ms, two additional 12-lead ECGs should be obtained over a brief period (e.g., 30 minutes) to confirm the finding. Patients are only eligible if a QTcF of <450ms is confirmed
10. Subjects must be ≥18 years of age.
11. Written informed consent obtained from the patient.
12. Both men and women enrolled in this trial must be in agreement with trial policy on contraception during the treatment phase of the study and 6 months afterwards. Egg donation, sperm donation and breastfeeding must be avoided.
13. Evidence of post-menopausal status or negative serum HCG pregnancy test for female pre menopausal patients. Women will be considered post-menopausal if they have been amenorrhoeic for 12 months without an alternative medical cause. The following age specific requirements apply:

    1. Women <50 years of age will be considered post-menopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinising hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilisation (bilateral oophorectomy or hysterectomy).
    2. Women ≥50 years of age will be considered post-menopausal if they have been amenorrhoeic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy induced menopause with last menses >1 year ago, or underwent surgical sterilisation (bilateral oophorectomy, bilateral salpingectomy, or hysterectomy).

Exclusion Criteria:

1. Previous diagnosis of RCC.
2. Metastatic or macroscopic residual disease.
3. Patients with positive resection margins after partial nephrectomy.
4. Patients with a single pulmonary nodule ≥5mm diameter are not eligible unless the nodule has had a definite benign diagnosis. Patients with multiple small, less than 5 mm nodules may be eligible if nodules have been shown to be radiologically stable for at least 8 weeks.
5. Prior anticancer treatment (other than nephrectomy) for RCC.
6. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

   1. Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
   2. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab or tremelimumab may be included only after consultation with the Study Physician.
7. History of another primary malignancy except for:

   1. Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence.
   2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
   3. Adequately treated carcinoma in situ without evidence of disease.
8. History of leptomeningeal carcinomatosis.
9. Concurrent enrolment in another clinical study, unless it is an observational (non interventional) clinical study or during the follow up period of an interventional study.
10. Major surgical procedure (as defined by the Investigator) within 28 days prior to the start of treatment. Local surgery of isolated lesions for palliative intent is acceptable.
11. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab or tremelimumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid.
12. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

    1. Patients with vitiligo or alopecia
    2. Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
    3. Any chronic skin condition that does not require systemic therapy
    4. Patients without active disease in the last 5 years may be included but only after consultation with the RAMPART Trial Management Team
    5. Patients with coeliac disease controlled by diet alone
13. A history of immunodeficiency syndrome. Please consult the MRC CTU at UCL on an individual basis if there is any uncertainty.
14. History of allogeneic organ transplant.
15. Uncontrolled intercurrent illness including, but not limited to:

    1. Ongoing or active infection of any kind (patients who are exhibiting symptoms consistent with COVID-19, or who have tested positive, should not be randomised into the study until they are asymptomatic and at least 14 days after a positive test)
    2. Symptomatic congestive heart failure
    3. Uncontrolled hypertension
    4. Unstable angina pectoris
    5. Uncontrolled cardiac arrhythmia
    6. Active peptic ulcer disease or gastritis
    7. Active bleeding diatheses
    8. Psychiatric illness or social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent.
16. Active infection including

    1. Tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice)
    2. Hepatitis B (known positive HBV surface antigen (HBsAg) result). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti HBc] and absence of HBsAg) are eligible.
    3. Hepatitis C
    4. Human immunodeficiency virus (positive HIV 1/2 antibodies). Note: Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
17. Receipt of live attenuated vaccine within 30 days prior to the start of treatment. Note: Patients, if enrolled, should not receive live vaccine while receiving investigational medicinal product and up to 30 days after the last dose of investigational medicinal product.
18. Pregnant or breastfeeding patients.
19. Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results.
20. Known allergy or hypersensitivity to durvalumab or tremelimumab, or any of their excipients.
21. Previous investigational medicinal product assignment in the present study.
22. Clinically significant pneumonitis or fibrosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1750 (Estimated)
Dates: Start 2018-07-19 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2034-12-01 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival (DFS): Arm C vs A | 6.25 years
  Interval from randomisation to first evidence of local recurrence, new primary RCC, distant metastases, or death from any cause, whichever occurs first.
Disease Free Survival (DFS): Arm B vs A | 10.54 years
  Interval from randomisation to first evidence of local recurrence, new primary RCC, distant metastases, or death from any cause, whichever occurs first.
Overall Survival (OS): Arm C vs A (high risk patients only) | 13.25 years
  All-cause mortality, the time from randomisation to death from any cause (including RCC).
Overall Survival (OS): Arm B vs A (high risk patients only) | 20.5 years
  All-cause mortality, the time from randomisation to death from any cause (including RCC).

SECONDARY OUTCOMES:
Metastasis-free survival (MFS): Arm C vs A | 6.25 years
  Interval from randomisation to first evidence of metastases or death from RCC
Metastasis-free survival (MFS): Arm B vs A | 10.54 years
  Interval from randomisation to first evidence of metastases or death from RCC
RCC specific survival time: Arm C vs A | 13.25 years
  Time from randomisation to death from RCC
RCC specific survival time: Arm C vs A | 20.5 years
  Time from randomisation to death from RCC

CONTACTS AND LOCATIONS:
Overall Officials: James Larkin, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (35):
- United Kingdom (35):
  - Aberdeen Royal Infirmary, Aberdeen
  - Ysbyty Gwynedd, Bangor
  - Royal Bournemouth Hospital, Bournemouth
  - Bristol Haematology and Oncology Centre, Bristol
  - Addenbrookes Hospital, Cambridge
  - Velindre Cancer Centre, Cardiff
  - Broomfield Hospital, Chelmsford
  - Cheltenham General Hospital, Cheltenham
  - Colchester General Hospital, Colchester
  - University Hospital Coventry & Warwickshire, Coventry
  - Western General Hospital, Edinburgh
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Diana Princess of Wales Hospital, Grimsby
  - Castle Hill Hospital, Hull
  - Raigmore Hospital, Inverness
  - St James University Hospital, Leeds
  - Leicester Royal Infirmary, Leicester
  - Clatterbridge Cancer Centre, Liverpool
  - St Bartholomew's Hospital, London
  - Mount Vernon Hospital, London
  - Royal Free Hospital, London
  - Guy's Hospital, London
  - Royal Marsden Hospital, London
  - Charing Cross Hospital, London
  - The Christie, Manchester
  - Nottingham University Hospital, Nottingham
  - Churchill Hospital, Oxford
  - Glan Clwyd Hospital, Rhyl
  - Scunthorpe General Hospital, Scunthorpe
  - Weston Park Hospital, Sheffield
  - South Tyneside District Hospital, South Shields
  - Southend University Hospital, Southend-on-Sea
  - Sunderland Royal Hospital, Sunderland
  - Royal Marsden Hospital, Sutton
  - Torbay Hospital, Torquay

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Oza B, Frangou E, Smith B, Bryant H, Kaplan R, Choodari-Oskooei B, Powles T, Stewart GD, Albiges L, Bex A, Choueiri TK, Davis ID, Eisen T, Fielding A, Harrison D, McWhirter A, Mulhere S, Nathan P, Rini B, Ritchie A, Scovell S, Shakeshaft C, Stockler MR, Thorogood N, Parmar MKB, Larkin J, Meade A. RAMPART: A phase III multi-arm multi-stage trial of adjuvant checkpoint inhibitors in patients with resected primary renal cell carcinoma (RCC) at high or intermediate risk of relapse. Contemp Clin Trials. 2021 Sep;108:106482. doi: 10.1016/j.cct.2021.106482. Epub 2021 Sep 16. PMID 34538402
- [Derived] Meade A, Oza B, Frangou E, Smith B, Bryant H, Kaplan R, Choodari-Oskooei B, Powles T, Stewart GD, Albiges L, Bex A, Choueiri TK, Davis ID, Eisen T, Fielding A, Harrison DJ, McWhirter A, Mulhere S, Nathan P, Rini B, Ritchie A, Scovell S, Shakeshaft C, Stockler MR, Thorogood N, Larkin J, Parmar MKB. RAMPART: A model for a regulatory-ready academic-led phase III trial in the adjuvant renal cell carcinoma setting. Contemp Clin Trials. 2021 Sep;108:106481. doi: 10.1016/j.cct.2021.106481. Epub 2021 Sep 16. PMID 34538401
- [Derived] Marconi L, Sun M, Beisland C, Klatte T, Ljungberg B, Stewart GD, Dabestani S, Choueiri TK, Bex A. Prevalence, Disease-free, and Overall Survival of Contemporary Patients With Renal Cell Carcinoma Eligible for Adjuvant Checkpoint Inhibitor Trials. Clin Genitourin Cancer. 2021 Apr;19(2):e92-e99. doi: 10.1016/j.clgc.2020.12.005. Epub 2021 Jan 7. PMID 33526329